CLINICAL TRIAL: NCT02379377
Title: PET Imaging of Hepatocellular Carcinoma With 18F-FSPG
Brief Title: 18F-FSPG PET in Imaging Patients With Liver Cancer Before Undergoing Surgery or Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1084; NCI-2015-00184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U24CA220325 (NIH)
Record Dates: First submitted 2015-02-06; First posted 2015-03-04 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Adult Hepatocellular Carcinoma; Resectable Hepatocellular Carcinoma; Cholangiocarcinoma; Benign Liver Tumor; Metastases to Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — carbon-11 acetate; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Cohorts A and B are Parallel. Cohorts C and D are Single Group. Cohorts E and F Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diagnostic (18F-FSPG PET) (Experimental): Patients undergo an 18F-FSPG PET scan within 4 weeks of surgery or OLT. Patients may also receive a second 18F-FSPG PET scan following standard-of-care treatment.
  Interventions: Biological: Fluorine F 18 L-glutamate Derivative 18F-FSPG; Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis
- Diagnostic (11C-Acetate PET or 18F-FDG PET) (Experimental): Patients may undergo either carbon-11 (11C)-Acetate PET or 18F-FDG PET scans within 4 weeks of surgery or OLT.
  Interventions: Biological: Fluorine F 18 L-glutamate Derivative 18F-FSPG; Biological: Carbon C 11 Acetate; Procedure: Positron Emission Tomography; Other: Laboratory Biomarker Analysis; Biological: Fluorine F 18 2-deoxy-2-(18F)fluoro-D-glucose

INTERVENTIONS:
Biological: Fluorine F 18 L-glutamate Derivative 18F-FSPG — Undergo 18F-FSPG PET scan
  Other Names: BAY94-9392
Biological: Carbon C 11 Acetate — Undergo 11C-acetate PET scan
  Other Names: 11C-acetate
  Arms: Diagnostic (11C-Acetate PET or 18F-FDG PET)
Procedure: Positron Emission Tomography — Undergo 18F-FSPG, 11C-acetate, or 18F-FDG PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Fluorine F 18 2-deoxy-2-(18F)fluoro-D-glucose — Undergo 18F-FDG PET scan
  Other Names: 18F-FDG
  Arms: Diagnostic (11C-Acetate PET or 18F-FDG PET)

SUMMARY:
This clinical trial studies fluorine F 18 L-glutamate derivative BAY94-9392 (18F-FSPG) positron emission tomography (PET) in imaging patients with liver cancer before undergoing surgery or transplant. Diagnostic procedures, such as 18F-FSPG PET, may help find and diagnose liver cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the relationship between 18F-FSPG PET/computed tomography (CT), pathology, and cancer metabolism in patients with suspected hepatocellular carcinoma (HCC) scheduled for liver resection surgery and orthotopic liver transplant (OLT).

II. To compare 18F-FSPG PET/CT with standard-of-care (SOC) diagnostic MRI imaging in patients with suspected HCC scheduled for liver resection surgery or OLT.

III. To compare the uptake of 18F-FSPG PET/CT with 11C-acetate PET/CT AND 18F-FDG PET/CT in suspected HCC and background liver in patients scheduled for liver resection surgery or OLT.

IV. To evaluate uptake of 18F-FSPG PET/CT in benign liver lesions compared to background.

V. To evaluate uptake of 18F-FSPG PET/CT in malignant non-HCC liver tumors.

OUTLINE:

Patients undergo 18F-FSPG PET and either carbon-11 (11C)-acetate PET or 18F-FDG PET scans within 4 weeks of surgery or OLT.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC with one or more of the following:

   1. Liver mass with non-rim arterial phase hyperenhancement (APHE) and one of the following: 1) 10-19 mm with ≥2 additional major features according to LI-RADS criteria ("washout", enhancing "capsule", and/or threshold growth), 2) 10-19 mm with "washout" and visibility at antecedent ultrasound (US) but with no "capsule" or threshold growth, 3) 10-19 mm with ≥50% size increase in ≤6 months but with no "washout" or "capsule" or 4) ≥20 mm with ≥1 additional major feature according to LI-RADS criteria ("washout", enhancing "capsule", or threshold growth).
   2. Lesions that meet LI-RADS 4 criteria or
   3. Lesions that meet LI-RADS 5 criteria or
   4. Suggestive imaging findings plus AFP > 200 mg/dL or
   5. Tumor confirmed by arteriography or
   6. Pathologic confirmation of tumor or
2. Diagnosis of a benign abdominal or pelvic tumor with the following characteristics:

   1. Liver mass (≥ 1 cm) that has suggestive imaging findings of a benign liver mass (adenoma, hemangioma, focal nodular hyperplasia).
   2. Prior SOC MRI or CT of the benign lesion within 8 weeks of enrollment or
3. Diagnosis of a malignant non-HCC liver tumor with one or more of the following characteristics:

   1. Liver mass (≥ 1 cm) that is biopsy proven, MRI-confirmed, or CT-confirmed metastatic disease (metastatic colorectal cancer, metastatic pancreatic cancer).
   2. Liver mass (≥ 1 cm) that is a non-HCC primary malignancy (cholangiocarcinoma).
   3. Prior SOC MRI or CT of the malignant non-HCC liver tumor within 8 weeks of enrollment or
4. Diagnosis of oligometastatic solid tumors in the following disease sites: colorectal, sarcoma, lung, head and neck, ovarian, renal, melanoma, pancreatic, prostate, cervix, breast, uterine and cholangiocarcinoma undergoing local consolidative therapy.

   and
5. Each patient must have completed conventional imaging and staging and MRI or CT before initiation of the investigational PET studies.

   and
6. Participants with HCC must be a candidate for liver resection, orthotopic liver transplant (OLT), or Y90 radioembolization.

Exclusion Criteria:

1. Participants under the age of 18 will be excluded from this study.
2. Participants who have HCC or cholangiocarcinoma but are not candidates for liver resection surgery or OLT, or Y90 radioembolization.
3. Pregnant and breastfeeding patients. Adequate birth control measures (oral, implanted, or barrier methods) must be used by all female participants of childbearing potential until all research PET scans are completed. Female participants of childbearing potential must have a negative serum or urine pregnancy test within 24 hours of the proposed investigational PET/CT scan(s) prior to injection of the investigational radiopharmaceutical.
4. Participants with poorly controlled diabetes mellitus (fasting blood glucose level > 200 mg/dL).
5. Participants with a known Infiltrative variant of HCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
18F-FSPG PET standardized uptake value (SUV) | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  The Standardized Uptake Value (SUV) for 18F-FSPG PET images will be determined in the hepatocellular carcinoma (HCC) tumor lesions, non-HCC liver tumors (benign), and background liver (normal tissue). These metrics include SUVmax, SUVpeak, or SUVmean and are common PET imaging measures.
11C-acetate standardized uptake value (SUV) | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  The Standardized Uptake Value (SUV) for 11C-acetate PET images will be determined in the tumor lesions and background liver (normal tissue). These metrics include SUVmax, SUVpeak, or SUVmean and are common PET imaging measures.
18F-FDG standardized uptake value (SUV) | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  The Standardized Uptake Value (SUV) for 18F-FDG PET images will be determined in the hepatocellular carcinoma (HCC) tumor lesions and background liver (normal tissue). These metrics include SUVmax, SUVpeak, or SUVmean and are common PET imaging measures.
Pharmacokinetics of 18F-FSPG, 11C-acetate, and 18F-FDG | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  The pharmacokinetics of 18F-FSPG, 11C-acetate and 18F-FDG uptake will be determined using compartmental modeling of PET imaging data. Venous samples will be collected over the course of 18F-FSPG, 11C-acetate and 18F-FDG scans to confirm blood pool radioactivity, evaluate metabolism, and to calibrate image-derived input functions. We will also utilize blood samples collected prior to scanning to assay plasma levels of carbon-12 acetate and glucose in each patient to explore normalizing pharmacokinetic parameters across patients.
Number of lesions | Within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  The number of lesions detected by 18F-FSPG PET will be determined and compared to the number of lesions detected by standard-of-care MRI, 11C-acetate PET, or 18F-FDG PET on a per patient basis.
Sensitivity of 18F-FSPG PET imaging | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  Sensitivity is defined as the true positive rate. It is defined as true positive/(true positive + false negative). The determination of HCC status will be based on diagnostic pathology.
Specificity of 18F-FSPG PET imaging | Within 4 weeks of standard-of-care imaging, within 4 weeks of liver resection surgery, within 12 months of orthotopic liver transplant and prior to therapy
  Specificity is defined as the true negative rate. It is defined as true negative/(true negative + false positive). The determination of HCC status will be based on diagnostic pathology.
Diagnostic pathology | After surgery; Through study completion, up to 4 years
  Tissue samples will be obtained for patients following either liver resection surgery or orthotopic liver transplant. Pathology will be performed on these tumor tissues as the gold-standard assessment to confirm the presence of HCC tumor. Histology will be correlated to PET imaging data.
Tumor grade | After surgery; Through study completion, up to 4 years
  Tissue samples will be obtained for patients following either liver resection surgery or orthotopic liver transplant. Tumor grade will be determined from pathology of tissue samples and correlated to PET imaging data for 18F-FSPG, 11C-acetate and 18F-FDG PET. The concordance of 18F-FSPG PET/CT and 11C-acetate PET/CT or 18F-FSPG PET/CT and 18F-FDG PET/CT will be evaluated. This will determine whether 18F-FSPG can be used singularly in place of combined use of 11C-acetate PET/CT (which typically detects low grade HCC) and 18F-FDG PET/CT (which typically detects high grade HCC).
Immunohistochemistry | After surgery; Through study completion, up to 4 years
  Tissue samples will be obtained for patients following liver resection surgery. The expression of immunohistochemical markers (ie. xC- and CD44) will be evaluated in these tumor tissues on an ordinal scale of 0, 1, 2 or 3 and correlated to 18F-FSPG PET imaging data. In addition, markers of inflammation and immune cell recruitment (ie. CD86, CD163, CD3), proliferation (Ki67), and apoptosis (Caspase 3) will also be evaluated and correlated to 18F-FSPG PET imaging data.

SECONDARY OUTCOMES:
Metabolic profile | After surgery; Through study completion, up to 4 years
  HCC tumor and non-cancerous liver tissue samples will be obtained for patients following liver resection surgery. Overall, tumoral tissue, peritumoral tissue and grossly normal surrounding liver will be evaluated. Metabolic profiles will be analyzed by mass spectrometry. The unbiased metabolomic phenome will be determined and correlated to 18F-FSPG PET.
Milan classification | Baseline prior to imaging and surgery
  Milan criteria will be applied to standard-of-care (SOC) MRI images. The number and size of lesions will be determined. A patient will be deemed to meet Milan criteria if they exhibit A) A single lesion 2 to 5 cm in diameter or B) Three or fewer tumors, each measuring 1 to 3 cm in diameter, and C) No evidence of extrahepatic involvement or microvascular invasion. The proportion of patients whose Milan classification by novel imaging classification changed following validation by histological confirmation will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Simone S Krebs, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org